CLINICAL TRIAL: NCT01378962
Title: Phase II, Open-label Study of Erlotinib (Tarceva®) Treatment in Patients With Locally Advanced or Metastatic Non-small-cell Lung Cancer Who Present Activating Mutations in the Tyrosine Kinase Domain of the Epidermal Growth Factor Receptor (EGFR) - (TRIGGER)
Brief Title: A Study of Tarceva (Erlotinib) in Patients With Locally Advanced or Metastatic Non-Small Cell Lung Cancer (TRIGGER)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML25514
Record Dates: First submitted 2011-06-21; First posted 2011-06-23 (Estimated); Results first posted 2015-10-29 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2017-12

CONDITIONS: Non-Squamous Non-Small Cell Lung Cancer
MeSH Terms: interventions — Erlotinib Hydrochloride

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: erlotinib

INTERVENTIONS:
Drug: erlotinib — 150 mg orally once a day for 12 months
  Other Names: Tarceva

SUMMARY:
This single-arm, open-label study evaluated the efficacy and safety of Tarceva (erlotinib) in participants with locally advanced or metastatic non-small cell lung cancer. Participants received daily oral doses of 150 mg Tarceva. The anticipated time on study treatment was 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/=18 years of age
* Locally advanced or metastatic non-small cell lung cancer
* Measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST)
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Life expectancy over >/=12 weeks
* Adequate hematological, liver, or kidney function

Exclusion Criteria:

* Previous therapy against epidermal growth factor receptor for metastatic disease
* Treatment with investigational drug during the 3 weeks before enrollment
* History of neoplasm
* Patients with symptomatic cerebral metastases
* Unstable systemic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-03-31 (Actual); Primary Completion 2013-06-30 (Actual); Study Completion 2017-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (10):
- Italy (10):
  - IRCCS Istituto Nazionale Tumori Fondazione Pascale; Oncologia Medica A, Napoli, Campania
  - Ospedale Bellaria; U.O. Oncologia Medica, Bologna, Emilia-Romagna
  - A.O. Universitaria Policlinico Di Modena; Ematologia, Modena, Emilia-Romagna
  - Istituto Regina Elena; Oncologia Medica A, Rome, Lazio
  - Istituto Europeo Di Oncologia, Milan, Lombardy
  - Istituto Clinico Humanitas;U.O. Oncologia Medica Ed Ematologia, Rozzano, Lombardy
  - Az Ospedaliera Nuovo Garibaldi Quartiere Nesima; Oncologia Medica, Catania, Sicily
  - Policlinico P. Giaccone; Istituto Di Oncologia, Clinica Medica 1, Palermo, Sicily
  - A.O. Universitaria Pisana-Ospedale Cisanello; Dipartimento Cardio Toracico-Pneumologia Ii, Pisa, Tuscany
  - Azienda Ospedaliera Di Perugia Ospedale s. Maria Della Misericordia; Oncologia Medica, Perugia, Umbria

RESULTS

PARTICIPANT FLOW:
Groups:
- Erlotinib 150 mg: Erlotinib 150 milligrams (mg) tablet orally once daily up to end of study (12 months) or until disease progression, unacceptable toxicity or consent withdrawal.
Period: Overall Study
Arm/Group | Erlotinib 150 mg
Started | 50
Completed | 33
Not Completed | 17
Not completed — Death | 14
Not completed — Lost to Follow-up | 1
Not completed — Other | 2

BASELINE CHARACTERISTICS:
Population: Safety population included all participants enrolled in the study who received at least 1 dose of treatment and had at least 1 safety assessment.
Groups:
- Erlotinib 150 mg: Erlotinib 150 mg tablet orally once daily up to end of study (12 months) or until disease progression, unacceptable toxicity or consent withdrawal.
Arm/Group | Erlotinib 150 mg
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.86 (11.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 16

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Disease Progression or Death at 12 Months After Baseline
Description: According to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1), progressive disease (PD) was defined as at least a 20 percent (%) increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum of the longest diameter recorded since treatment started or the appearance of 1 or more new lesions. For non-target lesions, PD was defined as the appearance of 1 or more new lesions and/or unequivocal progression of existing non-target lesions.
Time Frame: 12 months
Population: Intent to treat (ITT) population included all participants enrolled in the study who received at least 1 dose of treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Erlotinib 150 mg
Number analyzed (Participants) | 50
percentage of participants | 42

2. Secondary Outcome: Percentage of Participants Who Died
Time Frame: Every 8 weeks during treatment, after discontinuation participants were followed for up to 1 year after enrollment of the last participant (maximum up to 27 months)
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Erlotinib 150 mg
Number analyzed (Participants) | 50
percentage of participants | 28

3. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization to the date of death due to any cause. OS was assessed using Kaplan-Meier method.
Time Frame: as for outcome 2
Population: ITT population.
Measure: Mean (Standard Error); unit: months
Arm/Group | Erlotinib 150 mg
Number analyzed (Participants) | 50
months | 17.48 (1.09)

4. Secondary Outcome: Percentage of Participants With a Response by Best Overall Response
Description: Tumor response was assessed according to RECIST v1.1. Complete response (CR): complete disappearance of all target lesions and non-target disease, with the exception of nodal disease. All nodes must decrease to normal (short axis less than 10 mm), with no new lesions. Partial response (PR): greater than or equal to (>=) 30% decrease under baseline of the sum of diameters of all target lesions. The short axis was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. No unequivocal progression of non-target disease, and no new lesions. PD: >=20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum of the longest diameter recorded since treatment started or the appearance of 1 or more new lesions. For non-target lesions, appearance of 1 or more new lesions and/or unequivocal progression of existing non-target lesions. Stable disease (SD): not qualifying for CR, PR, or PD.
Time Frame: Baseline up to disease progression or end of study (up to 12 Months)
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Erlotinib 150 mg
Number analyzed (Participants) | 50
percentage of participants
  CR | 6
  PR | 62
  SD | 12
  PD | 4
  Not estimated | 16

5. Secondary Outcome: Percentage of Participants With Objective Response
Description: Objective response was defined as the percentage of participants with CR or PR as best overall response by RECIST v1.1. To be assigned the status of PR or CR, changes in tumor measurements were to be confirmed by repeated assessments no less than 4 weeks after the criteria for response were first met. CR was defined as complete disappearance of all target lesions and non-target disease, with exception of nodal disease. All nodes, both target and non-target, must decrease to normal (short axis less than 10 mm), with no new lesions. PR was defined as >=30% decrease under baseline of sum of diameters of all target lesions. The short axis was used in sum for target nodes, while longest diameter was used in sum for all other target lesions. No unequivocal progression of non-target disease, and no new lesions. Participants with no tumor assessment after start of study treatment were considered as non-responders. The percentage of participants with response is presented.
Time Frame: Baseline up to disease progression or end of study (up to 12 Months)
Population: ITT population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Erlotinib 150 mg
Number analyzed (Participants) | 50
percentage of participants | 68 [53 to 80]

6. Primary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the time from baseline to the date of first occurrence of disease progression or death. According to RECIST v1.1, PD was defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum of the longest diameter recorded since treatment started or the appearance of 1 or more new lesions. For non-target lesions, PD was defined as the appearance of 1 or more new lesions and/or unequivocal progression of existing non-target lesions. PFS was assessed using Kaplan-Meier method.
Time Frame: Up to 1 year after enrollment of the last participant (maximum up to 27 months)
Population: ITT population.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Erlotinib 150 mg
Number analyzed (Participants) | 50
months | 12.58 [10.25 to 16.95]

7. Primary Outcome: Probability of Being Progression Free 12 Months After Baseline
Description: According to RECIST v1.1, PD was defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum of the longest diameter recorded since treatment started or the appearance of 1 or more new lesions. For non-target lesions, PD was defined as the appearance of 1 or more new lesions and/or unequivocal progression of existing non-target lesions.
Time Frame: 12 months
Population: ITT population.
Measure: Mean (Standard Error); unit: probability of being progression-free
Arm/Group | Erlotinib 150 mg
Number analyzed (Participants) | 50
probability of being progression-free | 0.51 (0.08)

8. Secondary Outcome: Percentage of Participants Achieving CR, PR, or SD as Best Overall Response
Description: The Disease Control Rate was defined as the percentage of participants who had CR or PR or SD as Best Overall Response achieved within the time between the first drug administration and documented disease progression or end of study. According to RECIST v1.1, CR was defined as complete disappearance of all target lesions and non-target disease, with the exception of nodal disease. All nodes, both target and non-target, must decrease to normal (short axis less than 10 mm), with no new lesions. PR was defined as >=30% decrease under baseline of the sum of diameters of all target lesions. The short axis was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. No unequivocal progression of non-target disease, and no new lesions. SD was defined as not qualifying for CR, PR, or PD.
Time Frame: Baseline up to disease progression or end of study (up to 12 Months)
Population: ITT population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Erlotinib 150 mg
Number analyzed (Participants) | 50
percentage of participants | 80 [66 to 90]

9. Secondary Outcome: Percentage of Participants With Primary and Secondary Resistance
Description: Primary resistance: participants did not reach SD or PR or CR before going to PD. Secondary resistance: participants experienced PD after having reached SD or PR or CR at least once. CR: complete disappearance of all target lesions and non-target disease, with the exception of nodal disease. All nodes must decrease to normal (short axis less than 10 mm), with no new lesions. PR: >=30% decrease under baseline of the sum of diameters of all target lesions. The short axis was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. No unequivocal progression of non-target disease, and no new lesions. PD: >=20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum of the longest diameter recorded since treatment started or the appearance of 1 or more new lesions. For non-target lesions, appearance of 1 or more new lesions and/or unequivocal progression of existing non-target lesions.
Time Frame: Baseline up to disease progression (up to 12 Months)
Population: Analysis population included all participants enrolled in the study who received at least 1 dose of treatment and who had a documented PD response during the study period.
Measure: Number; unit: percentage of participants
Arm/Group | Erlotinib 150 mg
Number analyzed (Participants) | 24
percentage of participants
  Primary resistance | 8.33
  Secondary resistance | 91.67

10. Secondary Outcome: Percentage of Participants With Epidermal Growth Factor Receptor (EGFR) Mutation by Mutation Type
Description: EGFR is a gene in the tumor tissues and mutations in this gene have been linked to a variety of tumors. Presence or absence of EGFR mutation was determined in liquid biopsies by reverse transcriptase-polymerase chain reaction (RT-PCR /Cobas).
Time Frame: Baseline, At progression of disease (up to 12 Months)
Population: Analysis population included all participants enrolled in the study who received at least 1 dose of treatment and who had samples for EGFR mutation. Here, 'N' (number of participants analyzed) signifies the number of participants analyzed for this outcome measure and 'n' signifies the number of participants analyzed at specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | Erlotinib 150 mg
Number analyzed (Participants) | 45
percentage of participants
  Baseline: EGFR18 Mutation (n=45) | 0.00
  Baseline: EGFR19 Codon Deletion Mutation (n=45) | 51.11
  Baseline: EGFR20 Codon T790M Mutation (n=45) | 2.22
  Baseline: EGFR21 Codon L585R Mutation (n=45) | 15.56
  At PD: EGFR18 Mutation (n=18) | 0.00
  At PD: EGFR19 Codon Deletion Mutation (n=18) | 50.00
  At PD: EGFR20 Codon T790M Mutation (n=18) | 27.78
  At PD: EGFR21 Codon L585R Mutation (n=18) | 16.67

ADVERSE EVENTS:
Time Frame: Up to 1 year after enrollment of the last participant (maximum up to 27 months)
Description: Safety population included all participants enrolled in the study who received at least one dose of treatment and had at least one safety assessment.
Arm/Group | Erlotinib 150 mg
Serious Adverse Events (participants affected / at risk) | 10/50
Other Adverse Events (participants affected / at risk) | 46/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib 150 mg (N=50)
Cardiac failure acute (Cardiac disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 1
Pneumonia (Infections and infestations) | 2
Hip fracture (Injury, poisoning and procedural complications) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Convulsion (Nervous system disorders) | 1
Hemiplegia (Nervous system disorders) | 1
Confusional state (Psychiatric disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Jugular vein thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib 150 mg (N=50)
Vertigo (Ear and labyrinth disorders) | 4
Conjunctivitis (Eye disorders) | 11
Abdominal pain upper (Gastrointestinal disorders) | 4
Diarrhoea (Gastrointestinal disorders) | 27
Stomatitis (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 4
Asthenia (General disorders) | 9
Chest pain (General disorders) | 7
Fatigue (General disorders) | 5
Pyrexia (General disorders) | 9
Paronychia (Infections and infestations) | 7
Contrast media reaction (Injury, poisoning and procedural complications) | 3
Blood bilirubin increased (Investigations) | 3
Decreased appetite (Metabolism and nutrition disorders) | 6
Back pain (Musculoskeletal and connective tissue disorders) | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 10
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4
Alopecia (Skin and subcutaneous tissue disorders) | 7
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 5
Dry skin (Skin and subcutaneous tissue disorders) | 4
Pruritus (Skin and subcutaneous tissue disorders) | 10
Rash (Skin and subcutaneous tissue disorders) | 36
Skin ulcer (Skin and subcutaneous tissue disorders) | 4
Nausea (Gastrointestinal disorders) | 3
Oedema peripheral (General disorders) | 3
Cystitis (Infections and infestations) | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3
Nail disorder (Skin and subcutaneous tissue disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.